CLINICAL TRIAL: NCT00914303
Title: A Phase I, Single Centre, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability and Pharmacokinetics of Extended Release Tablets of AZD3241 After Administration of Multiple Ascending Doses in Healthy Male and Female Volunteers Including Food Effect
Brief Title: Study to Evaluate Different Extended Release (ER)-Formulations and Multiple Ascending Dosing of AZD3241
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Rolf Karlsten , MD, PhD, Medical Science Director, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D0490C00002; EudraCT No 2007-003145-33
Record Dates: First submitted 2009-06-01; First posted 2009-06-04 (Estimated); Last update posted 2010-04-06 (Estimated); Status verified 2010-04

CONDITIONS: Healthy
Keywords: Safety; tolerability; healthy; Healthy volunteer study
MeSH Terms: interventions — AZD3241

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AZD3241 (Experimental): AZD3241 Tablets
  Interventions: Drug: AZD3241
- Placebo (Experimental): Placebo Tablets
  Interventions: Drug: Placebo Tablet

INTERVENTIONS:
Drug: AZD3241 — Oral Tablet, Repeated Administration
  Arms: AZD3241
Drug: Placebo Tablet — Oral Tablet. Repeated Administration
  Arms: Placebo

SUMMARY:
The aims of the study are to assess the safety, tolerability and pharmacokinetics of ER tablets of AZD3241 following multiple ascending doses administered to healthy male and female subjects including the effect of food.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects 30-65 years
* Body Mass Index (BMI) between 18 and 30 kg/m2 and weigh at least 50 kg and no more than 100 kg

Exclusion Criteria:

* History of any clinically significant disease or disorder
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
* Previous history of frequent pre-syncope or syncope

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2009-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Safety variables (adverse events, vital signs, ECG, safety lab) | Assessments performed at frequent timepoints during a 4-8 week period

SECONDARY OUTCOMES:
To characterize the pharmacokinetics of AZD3241 in plasma | Frequent sampling occasions during some study days for a 4-8 weeks period

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Karlsten, MD, Study Director — Medical Science Director AstraZeneca R&D Södertälje.; Wolfgang Kuhn, MD, PhD, Principal Investigator — Quintiles AB Phase I Unit, Uppsala, Sweden
Locations (1):
- Research Site, Uppsala, Sweden